CLINICAL TRIAL: NCT02357745
Title: Biochemical Evaluation of Plasma,Urine and Salivary Neopterin Levels in Pre and Post-menopausal Women With Periodontitis Following Non-surgical Therapy
Brief Title: Evaluation of Neopterin Levels in Pre and Post-menopausal Women With Periodontitis Following Non Surgical Therapy
Acronym: ENLPPMNS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, DR.CH.SUMADHURA, SUMADHURA, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Other Study IDs: suma thesis
Record Dates: First submitted 2015-01-21; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Periodontitis
Keywords: neopterin; plasma; urine; saliva; menopause; periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre-menopausal with periodontitis: non surgical periodontal therapy ( scaling and root planing)
  Interventions: Procedure: Non surgical periodontal therapy
- Post-menopausal with periodontitis: non surgical periodontal therapy ( scaling and root planing)
  Interventions: Procedure: Non surgical periodontal therapy

INTERVENTIONS:
Procedure: Non surgical periodontal therapy — scaling and root planing

SUMMARY:
Neopterin has been identified as a marker of cellular immune system activation. It is synthesized by macrophages upon stimulation with the cytokine interferon-gamma and is indicative of a pro-inflammatory immune status. Neopterin concentration increases with increasing severity of periodontal disease in diverse body fluids like Urine, Saliva and Plasma. Hence Neopterin can be considered as an important inflammatory marker in periodontal disease as well as other systemic diseases.

DETAILED DESCRIPTION:
At baseline - plasma, urine and saliva samples were collected and analysed for neopterin levels from the pre and post-menopausal women with periodontitis . Followed by scaling and root planing done in both the groups. After 3 months again these 3 samples were collected and analysed for post treatment neopterin levels

ELIGIBILITY:
Inclusion Criteria:

* moderate to chronic periodontitis
* non-smokers
* minimum 15 natural teeth present

Exclusion Criteria:

* patients on long term steroid medication
* with gross oral pathology or tumors
* undergoing hormone replacement therapy
* not undergone periodontal therapy in past 6 months
* under medication in past 6 months
* systemic disorders and drugs which influence the periodontium

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 15 pre-menopausal women with periodontitis 15 post-menopausal women with periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Co-relating neopterin and periodontitis levels in pre and post menopausal women | 3 months

REFERENCES:
- [Background] Bakhtadze MG, Margvelashvili VV, Kamkamidze GK. [Interferon-gamma and neopterin in blood serum of patients with chronic periodontitis after autograft operations]. Georgian Med News. 2006 Mar;(132):30-3. Russian. PMID 16636374
- [Result] Arjunkumar R, Sudhakar U, Jayakumar P, Arunachalam L, Suresh S, Virupapuram P. Comparative analysis of gingival crevicular fluid neopterin levels in health and periodontal disease: a biochemical study. Indian J Dent Res. 2013 Sep-Oct;24(5):582-6. doi: 10.4103/0970-9290.123376. PMID 24355959
- [Result] Pradeep AR, Kumar MS, Ramachandraprasad MV, Shikha C. Gingival crevicular fluid levels of neopterin in healthy subjects and in patients with different periodontal diseases. J Periodontol. 2007 Oct;78(10):1962-7. doi: 10.1902/jop.2007.070096. PMID 18062118
- [Result] Ozmeric N, Baydar T, Bodur A, Engin AB, Uraz A, Eren K, Sahin G. Level of neopterin, a marker of immune cell activation in gingival crevicular fluid, saliva, and urine in patients with aggressive periodontitis. J Periodontol. 2002 Jul;73(7):720-5. doi: 10.1902/jop.2002.73.7.720. PMID 12146530
- [Result] Vrecko K, Staedtler P, Mischak I, Maresch L, Reibnegger G. Periodontitis and concentrations of the cellular immune activation marker neopterin in saliva and urine. Clin Chim Acta. 1997 Dec 10;268(1-2):31-40. doi: 10.1016/s0009-8981(97)00154-x. PMID 9495569
- [Result] Bakhtadze MG, Margvelashvili VV, Kamkamidze GK. [Interferon-gamma and neopterin in blood serum of patients with chronic periodontitis]. Georgian Med News. 2006 Jan;(130):50-3. Russian. PMID 16510912